CLINICAL TRIAL: NCT01933711
Title: Rituximab Maintenance Therapy Versus Observation in Aggressive CD20+ Lymphoma and Mantle Cell Lymphoma - a Prospective Randomized Phase III Trial
Brief Title: Rituximab Maintenance Therapy in Aggressive CD20 (Cluster of Differentiation Antigen 20) Positive Lymphoma and Mantle Cell Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Mathias Witzens-Harig, Priv.Doz Dr.med., University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD2002
Record Dates: First submitted 2013-08-23; First posted 2013-09-02 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: CD20+ Aggressive Lymphoma, Mantle Cell Lymphoma
Keywords: CD20+ aggressive lymphoma; mantle cell lymphoma; rituximab; maintenance
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rituximab maintenance (Experimental): maintenance therapy with rituximab (375 mg/m2) administered every 3 months for 2 years.
  Interventions: Drug: rituximab
- Observation (No Intervention): observational arm, no intervention

INTERVENTIONS:
Drug: rituximab
  Arms: Rituximab maintenance

SUMMARY:
Clinical and pharmacokinetic data suggest that the effect of rituximab could be improved by prolonged exposure to the drug. To test for this hypothesis we performed a prospective randomized trial of rituximab maintenance therapy versus observation in patients (pts) with aggressive CD20+ B-cell lymphoma and mantle cell lymphoma.

DETAILED DESCRIPTION:
After completion of standard treatment, pts with aggressive CD20+ B-cell lymphoma and mantle cell lymphoma were randomized to either observation or maintenance therapy with rituximab (375 mg/m2) administered every 3 months for 2 years. Both pts after first line therapy and pts after relapse treatment were included in the study. Pts with aggressive lymphoma were enrolled if they had achieved a complete response (CR) after initial treatment. Pts with aggressive lymphoma with residual tumor mass underwent positron emission tomography (PET) and qualified for randomization if this examination showed no signs of tumor activity. Pts with mantle cell lymphoma were eligible for the study if at least a partial response (PR) was achieved. Primary endpoint of the study was progression free survival (PFS), secondary endpoints were time to progression (TTP), overall survival (OS) and response to treatment. Differences between PFS and OS were analysed using the logrank test and the proportional hazard model of Cox. TTP was analyzed using a competing risk model with death as competing event.

ELIGIBILITY:
Inclusion Criteria:

* aggressive B-cell lymphoma or mantle cell lymphoma
* CR (complete remission) oder CRu (complete remission unconfirmed) after previous therapy
* PR (partial remission) only when PET is negative
* minimal age 18 years
* CD20+ expression on tumor cells
* effective contraception
* Karnofsky status > 60
* written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2002-07; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 24 months after randomization
  Primary endpoint of the study was progression free survival (PFS)

SECONDARY OUTCOMES:
time to progression (TTP) | 24 months after randomization
overall survival (OS) | 24 months after randomization
response to treatment | 24 months after randomization

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - University of Heidelberg Hospital, Heidelberg, Baden-Wurttemberg
  - University of Mannheim Hospital, Mannheim, Baden-Wurttemberg
  - University of Bonn Hospital, Bonn, Nordhein-Westfalen